CLINICAL TRIAL: NCT06834282
Title: Phase 1/1b First-in-human Study of Autologous Chimeric Engulfment Receptor T-Cell CER-1236 in Patients With Acute Myeloid Leukemia (CertainT-1)
Brief Title: CER-1236 in Patients With Acute Myeloid Leukemia (AML)
Acronym: CertainT-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CERo Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-1-1
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-02

CONDITIONS: AML; Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: Relapsed Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; Mesna

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose and dose expansion study of CER-1236 administered as a single agent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Agent CER-1236 (Experimental): AML patient treated with a single dose of CER-1236 monotherapy
  Interventions: Drug: CER-1236; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Part 2: Single Agent CER-1236 (Experimental): AML patient treated with a single dose of CER-1236 monotherapy
  Interventions: Drug: CER-1236; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna

INTERVENTIONS:
Drug: CER-1236 — an autologous chimeric engulfment receptor T-cell
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Mesna — Chemoprotectant

SUMMARY:
This is a ﬁrst in human, multi center, open label, phase 1/1b study to evaluate the safety and preliminary efﬁcacy of CER-1236 in patients with relapsed/refractory (R/R), measurable residual disease (MRD) positive acute myeloid leukemia (AML), or TP53mut disease.

DETAILED DESCRIPTION:
CER-1236 is a first in class chimeric engulfment receptor T-cell therapy candidate that targets the Tim4 ligand.

This is a ﬁrst in human, multi center, open label, phase 1/1b study to evaluate the safety and preliminary efﬁcacy of CER-1236 in patients with relapsed/refractory (R/R), measurable residual disease (MRD) positive acute myeloid leukemia (AML), or TP53mut disease.

The study is divided into Part 1 (escalation phase) and Part 2 (expansion phase).

Part 1 (Escalation Phase): The primary objectives of Part 1 are to deﬁne the safety of different doses of CER-1236 and to deﬁne the recommended dose for Part 2 (RP2D) of CER-1236.

Part 2 (Expansion Phase): The objective of the Part 2 expansion cohort is to evaluate the safety and efﬁcacy of CER-1236 in patients with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to have a confirmed diagnosis of de novo or secondary AML, or myelodysplastic syndrome (MDS)/AML with 10% to 19% blasts, per the International Consensus Classification 2022 or the WHO 2022 classification.
* Absolute lymphocyte count >0.3 x 109/L prior to apheresis.
* Eastern cooperative oncology group (ECOG) performance status 0 to 1.

Exclusion Criteria:

* Prior therapy with a permanently integrated, genetically modified cell product.
* No measurable leukemia on the screening bone marrow evaluation prior to any bridging therapy.
* Active autoimmune disease or history of autoimmune disease requiring treatment within the prior 2 years. Patients with history of autoimmune thyroiditis or type 1 diabetes well controlled on replacement regimen are eligible.
* A known hypersensitivity or severe allergy to fludarabine, cyclophosphamide, or study drug components or diluents.
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the physician.
* Primary immunodeficiency disorder.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Part 1) | 2 year
  Escalation Period
Incidence of dose-limiting toxicities (DLTs) of CER-1236 Monotherapy - (Part 1) | 28 days
  Escalation Period
Estimation of the objective response rate (ORR), complete response (CR), composite complete response (cCR), and measurable residual disease (MRD) negativity rates - (Part 2) | 2 years
  Expansion Period

SECONDARY OUTCOMES:
Estimation of the objective response rate (ORR), complete response (CR), composite complete response (cCR), and measurable residual disease (MRD) negativity rates - (Part 1) | 2 years
  Escalation Period
PK (Cmax) of CER-1236 - (Part 1) | 2 years
  Escalation Period
PK (AUC) of CER-1236 - (Part 1) | 2 year
  Escalation Period
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Part 2) | 2 years
  Expansion Period

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Sarah Cannon Research Insitute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No